CLINICAL TRIAL: NCT01003626
Title: A Pilot Study Assessing the Feasibility and Safety of Measuring Interstitial Fluid Pressure (IFP) in Patients With Advanced Malignant Melanoma Before Starting Systemic Treatment
Brief Title: Interstitial Fluid Pressure (IFP) Pilot Study in Melanoma Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0120
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Advanced Cancers; Melanoma
Keywords: Advanced cutaneous melanoma; Tumor Pressure; Tumor IFP; Interstitial Fluid Pressure; IFP; Transducer-tipped catheter Mikro-Tip SPC-320; Transducer Millar; Power Lab 8/30 amplifier
MeSH Terms: conditions — Melanoma | interventions — Amplifiers, Electronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IFP Measurement (Experimental): Tumor interstitial fluid pressure (IFP) assessments
  Interventions: Procedure: Tumor Interstitial Fluid Pressure (IFP) assessments; Device: Transducer-catheter SPC-320 + Amplifier

INTERVENTIONS:
Procedure: Tumor Interstitial Fluid Pressure (IFP) assessments — The tip of a needle will be inserted in a skin lesion (similar to a biopsy needle) for up to 3 tumors. The needle is connected to a machine that reads the pressure inside the tumor. The whole process, including cleaning and numbing the lesion, will take about 3-4 minutes.
Device: Transducer-catheter SPC-320 + Amplifier — Transducer-tipped catheter Mikro-Tip SPC-320 and transducer Millar with Power Lab used to assess the interstitial fluid pressure in a malignant melanona nodule

SUMMARY:
The goal of this clinical research study is to learn about the side effects of measuring the tumor pressure in patients who have advanced melanoma and have not received chemotherapy. Researchers also want to learn if patients with a lower tumor pressure may respond better to chemotherapy.

DETAILED DESCRIPTION:
Tumor Pressure Testing:

If you are found to be eligible to take part in this study, the pressure in up to three tumors will be measured. Medical photography will also be used for documentation if needed.

This will be done in the melanoma outpatient clinic. You will be asked to lie down and the skin over the lesion will be cleaned with betadine (iodine) or a different cleaning agent if you are allergic to iodine. The skin over the lesion will then be numbed with anesthetic. A topical anesthetic is a local anesthetic that is used to numb the surface of a body part. Thirty minutes before the IFP measurement, an EMLA patch (Lidocaine 2.5% and Prilocaine 2.5%) will be applied on the surface of study. Your treating doctor may prescribe a pain drug to help with any discomfort the measurement may cause.

For the tumor measurement, the tip of a needle will be inserted in a skin lesion (similar to a biopsy needle). The needle is connected to a machine that reads the pressure inside the tumor. The measurement itself will take a few seconds. The whole process, including cleaning and numbing the lesion, will take about 3-4 minutes.

You will stay in the clinic and be monitored for side effects for about 1 hour following the tumor measurement.

At 3 days after the measurement, you will be asked if you have experienced any side effects. If you are not coming to the clinic, you will be called.

Length of Study:

You will be off study after you have completed two cycles of chemotherapy and the second set of tumor measurements are done.

Follow-Up:

After the 2 cycles of chemotherapy, you will be checked for tumor response. The IFP study will be finished at this time. You will also receive a phone call 30 days after the procedure to see if you have experienced any side effects.

This is an investigational study. Measuring tumor pressure before chemotherapy is investigational.

Up to 20 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologic confirmation of malignant melanoma and skin lesion, and/or subcutaneous metastases.
2. Males and Females >/= 18 years of age.
3. Subject is willing and able to comply with scheduled visits and other trial procedures.
4. Patients must be chemo-naive for malignant melanoma. Prior immunotherapy is allowed.
5. Must be scheduled for systemic chemotherapy within 3 weeks of measurements
6. Patient must have at least a one intact tumor or satellite lesion measuring >/= 10 mm in longest diameter.
7. Patients must sign and date an informed consent.

Exclusion Criteria:

1. Major surgery or radiation therapy close to the area where tumor IPF will be measured, within 4 weeks of starting the study treatment.
2. Patients with the only melanoma skin lesions being localized in the area of the head and neck.
3. High risk of bleeding with platelets </= 50,000 microliter, Partial thromboplastin time (PTT)/prothrombin time (PT) > 2 times upper limit of normal or patients on any type of anticoagulation.
4. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation, or may interfere with the interpretation of study results, and in the judgment of the investigator or his designee would make the subject inappropriate for entry into this study.
5. Patients will be excluded if they are receiving biological agents only.
6. Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Feasibility measured by proportion of patients in whom interstitial fluid pressure (IFP) can be measured | Baseline only + follow up 3 days after measurement

CONTACTS AND LOCATIONS:
Overall Officials: Jade Homsi, MD, Study Chair — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org